CLINICAL TRIAL: NCT03862066
Title: The Role of the Central Memory Phenotype in Predicting Response to PD-1 Inhibition in Pre-clinical Models of Oral Cancer
Brief Title: Memory Phenotype and PD-1 Inhibition Response in Oral Cancer
Status: Terminated | Type: Observational
Why Stopped: Low accrual progress per internal scientific review committee
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Other Study IDs: 102985
Record Dates: First submitted 2019-03-01; First posted 2019-03-05 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
Keywords: head and neck cancer
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms | interventions — Blood Specimen Collection; Tissue Banks

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue and blood specimens
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Received Nivolumab
  Interventions: Other: Blood collection; Other: Tissue collection
- Nivolumab Naive
  Interventions: Other: Blood collection; Other: Tissue collection

INTERVENTIONS:
Other: Blood collection — 5 milliliters (mL) of blood will be collected at the time of surgery
Other: Tissue collection — Left over tissue will be collected at the time of surgery

SUMMARY:
The purpose of this research study is collect tissue and blood samples from patients who are having surgery and use those samples in lab studies to see if there are any markers in blood and tissue that can help predict how cancer will react to different treatment. Participants in this study will have a blood sample and tissue samples collected for research. The blood and tissue collected will be tested in the laboratory. The tissue collected will be left over tissue from the standard of care surgery.

DETAILED DESCRIPTION:
Squamous cell carcinoma of the head and neck (HNSCC) is the sixth most common neoplasm in the world and despite advances in treatment, the 5-year survival remains approximately 50%. Because of the need for new therapies, the possibility of immunotherapeutic approaches for HNSCC patients has gained interest. Interest in this has continued as more than half of the subjects enrolled to an ongoing clinical trial in patients with with oral squamous cell carcinoma (OCSCC) have responded to neoadjuvant presurgical Nivolumab therapy. Additionally, unlike other solid tumors it appears responders have higher proportions of CD4+ tumor-infiltrating lymphocytes (TILs) whereas non-responders have an increase in CD8+ TILs population. Furthermore, the investigator's data suggests that response to PD-1 blockade is associated with an increase in CD45RA- CD62L+ population or central memory phenotype within TIL whereas progression of disease correlates with an increase in the CD45RA- CD62L- population or effector memory phenotype.

As previously demonstrated in several other tumor types the magnitude of response to immunotherapy directly correlates to presence of antigen specific T cells within the tumor and tumor microenvironment. Therefore, the long-term objective of this project is to identify predictive biomarkers of immune response from either TILs or tumor cells from patients with head and neck squamous carcinoma. To achieve this goal the overall objective of the current study is to develop a pre-clinical murine models in an effort to more completely evaluate the memory phenotype of TILs before and after PD-1 inhibition and to subsequently to determine the efficacy of TIL therapy in this mouse model of oral cancer. This project will test a central hypothesis that TILs derived from responders to neoadjuvant pre-surgical PD-1 inhibition in both a patient derived xenograft mouse model of oral cancer.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed histologically proven locoregional oral squamous cell carcinoma (OSCC) without evidence of distant metastases. OSCC includes the subsites of oral tongue, floor of mouth, gingiva, retromolar trigone and buccal mucosa OR

Recurrent or persistent histologically proven locoregional OSCC that was initially treated with surgery alone.

* must be eligible for surgical resection
* greater than 18 years of age

Exclusion Criteria:

* prior immunotherapy or treatment with another anti PD-1 agent besides nivolumab
* prior chemotherapy including cetuximab or radiation therapy
* concomitant malignancies except cutaneous squamous cell carcinoma or basal cell carcinoma
* unresectable primary tumor or regional disease or distant metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be selected from cancer patients being seen at MUSC.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2019-02-08 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-11-22 (Actual)

PRIMARY OUTCOMES:
Count of PDX models that are developed from patient samples | 6 months
  It is anticipated that there will be 12 successful PDX models developed as part of this study.

SECONDARY OUTCOMES:
Change in tumor growth in PDX models | 6 months
  Tumors will be measured with calipers bi-weekly and measurements will be plotted overtime.
Change in tumor volume in PDX models | 6 months
  Tumor volume with be calculated based on the two greatest dimensions of the tumor and will be plotted overtime.

CONTACTS AND LOCATIONS:
Overall Officials: David Neskey, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided